CLINICAL TRIAL: NCT02838641
Title: Application of GeneXpert on Bronchoscopic Samples for Patients Suspicious of TB
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, To Kin Wang, Honorary Clinical Assistant Professor, Chinese University of Hong Kong
Other Study IDs: 2014.556
Record Dates: First submitted 2016-07-18; First posted 2016-07-20 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Device: GeneXpert — Real time integrated and automated nucleic acid amplification test for detection of TB

SUMMARY:
This is an observational study using Bronchial-alveolar lavage (BAL) as specimen for GeneXpert, a real time polymerase chain reaction (PCR) test for detection of tuberculosis (TB). Patients suspicious of TB, who require bronchoscopy as part of the investigation procedures, will be recruited for this study over a period of 18 months. Clinical likelihood of TB will be systematically scored according to various clinical parameters. This will determine the pre-test probability. Clinician will decide if anti-TB treatment is to be started and patients will be followed up for a minimal of 18 months. Sensitivity, specificity, positive, negative predictive values and the respective likelihood ratio will be calculated accordingly.

ELIGIBILITY:
Inclusion Criteria:

1. Patients > 18 years old suspected of TB clinically.
2. Patients suspected of TB but both smear microscopy and TB PCR of sputum are negative or sputum cannot be produced.
3. BAL samples obtained following standard investigation procedure
4. CXR or CT imaging available.

Exclusion Criteria:

1. Bronchoscopy is not planned as a necessary procedure for investigation.
2. Diagnosis of active TB has been made by other means.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients suspected of TB but both smear microscopy and TB PCR of sputum are negative or sputum cannot be produced
Sampling Method: Non-Probability Sample
Enrollment: 219 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
sensitivity, specificity, positive and negative predictive values | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine and Therapeutics, Prince of Wales Hospital, CUHK, Shatin, Hong Kong